CLINICAL TRIAL: NCT05338658
Title: Phase I Study of Peptide Alarm Therapy (PAT) Administered by Intratumoral Injection With a PD-1/PD-L1 Inhibitor in Patients With Solid Tumor Cancers Who Have Failed 1 or More Prior Therapies
Brief Title: Study of PAT in Patients With Solid Tumor Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS105
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastasis; Solid Tumor
Keywords: PAT
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peptide Alarm Therapy + Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg every 3 weeks (Dose Finding Component) or a disease appropriate PD1/PD-L1 inhibitor (Dose Expansion Component) for 2 treatment courses per standard of care.
  The first dose of PAT is given on Day 1 and on Day 3 (36 to 48 hours after the 1st PAT dose)
  A second course of the PD1/PD-L1 inhibitor is given per standard of care on Day 22 (Cycle 2 Day 1).
  Interventions: Drug: Peptide Alarm Therapy (PAT)

INTERVENTIONS:
Drug: Peptide Alarm Therapy (PAT) — PAT is given on Day 1 by IT injection after the 1st anti PD-1/PD-L1 infusion and again 36-48 hours later on Day 3.
  Other Names: Pembrolizumab

SUMMARY:
This is a single center Phase I study with extension of peptide alarm therapy (PAT) administered by intratumoral (IT) injection during the 1st course of a standard of care intravenous PD-1/PD-L1 inhibitor for the treatment of locally advanced or metastatic solid tumor cancers that has failed to be controlled after one or more prior therapies including a previous PD-1/PD-L1 inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Must be seropositive for CMV and EBV.
* Must have at least one HLA-A*0201 allele. This screening can be performed after determining CMV and EBV seropositivity is established or, if available, from the results of previous tumor profiling by any CLIA-certified lab (i.e. Caris, FoundationOne).
* 18 years or older at the time of signing the pre-screening consent.
* ECOG Performance Status 0 or 1.
* Adequate organ function within 14 days of study enrollment
* Cardiac: New York Heart Association (NYHA) Functional Classification Class I.
* Pulmonary: oxygen saturation ≥ 90% on room air.
* Time between last dose of prior anti-cancer therapy and Day 1 of this study:

  * Chemotherapy: a minimum of 28 days since last treatment.
  * Targeted therapy, immunotherapy, investigational agents: a minimum of 45 days since last dose (at least 2 months for anti-VEGF)
  * Prior palliative radiotherapy within 7 days of start of study treatment. Participants must have recovered from all radiation-related toxicities (prior irradiation to targeted lesions is not permitted)
* Must have recovered to CTCAE ≤Grade 1 from previous treatment related acute toxicities.
* Persons of childbearing potential or with partners of childbearing potential must be willing to abstain from heterosexual activity or to use a highly effect form of contraception from the time of study enrollment until at least 4 months after the last dose of PD-1/PD-L1 inhibitor.
* Able to understand and provide voluntary written consent prior to the performance of any research related activity.

Exclusion Criteria:

* Pregnant or breast feeding.
* Requires therapeutic anticoagulation for which it is deemed unsafe to discontinue anticoagulation for 5 days prior to Cycle 1 through Day 7 of Cycle 1
* Class II or greater New York Heart Association Functional Classification criteria or serious cardiac arrhythmias likely to increase the risk of cardiac complications of therapy (e.g. ventricular tachycardia, frequent ventricular ectopy, or supraventricular tachyarrhythmia requiring chronic therapy)
* Known active CNS metastases
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to study enrollment.
* Prior bone marrow and/or solid organ transplant.
* Has severe hypersensitivity (≥Grade 3) to prior PD-1/PD-L1 and/or any of its excipients.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Known seropositive for HIV or known active Hepatitis B or C infection with detectable viral load by PCR
* Known history of active TB (Bacillus Tuberculosis)
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of peptide alarm therapy (PAT) | End of Treatment (typically at day 43)
  Use CTCAE v5 criteria to count toxicities per patient including proportions and their 95% confidence intervals will be calculated

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 Months
  Kaplan-Meier curves will be used to estimate with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No